CLINICAL TRIAL: NCT07123818
Title: AI for Detection of Brain Aneurysm: Low-cost Opportunistic Screening
Acronym: AIDALOS-III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Robovision BV (Industry); Universitair Ziekenhuis Brussel (Other); General Hospital Groeninge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Z-2025021
Record Dates: First submitted 2025-06-02; First posted 2025-08-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; Intracranial; UIA; Unruptured
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective multicentric interventional study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain NECT scans with possible UIA detected by AI software and radiologist (Other): Patients that have had a brain NECT scans on which the AI software detected a possible unruptured intracranial brain aneurysm (UIA) and which the radologist confirmed as possible UIA can participate in the study (= enrolled subjects). They are requested to sign Informed Consent Form (ICF) after which follow-up data regarding the untruptured intracranial aneurysm (UIA) will be gathered.
  Interventions: Device: AI software

INTERVENTIONS:
Device: AI software — AI software that will verify brain NECT scans on the presence of unruptured intracranial aneurysms (UIA). Brain NECT scans will be send to the AI software, after approval of the subject, which will detect possible unruptured intracranial aneurysms (UIA). NECT scans on which a possibe UIA has been detected will be transferred to a platform on which involved radiologist can verify the AI result(s).

SUMMARY:
The goal of this clinical trial is to verify the opportunistic screening potential of the AI software for detection of brain unruptured intracranial aneurysms (UIA) on routinely performed brain NECT scans in a prospective setting in the Belgian population.

The main question the study aims to answer is: Does the AI algorithm has potential to be used as clinical screening potential for detection of brain UIA on brain NECT scans?

The performance and the clinical use of the AI algorithm will be measured based on the number of UIA detected by the AI software compared to the number of UIA confirmed by review of a radiologist compared to the number of UIA already known by review of the electronic patient file/additional diagnostic research.

Participants will be followed-up following Standard-of-Care (SoC). In addition, participants will be requested to complete a questionnaire (the EQ-5D-5L questionnaire).

Furthermore, patient outcomes, complications/death related to the possible (un)ruptured brain aneurysm will be assessed 5 years after study enrolment.

ELIGIBILITY:
Inclusion Criteria:

* the subject of the NECT scan must be an adult patient (Age ≥ 18 years old);
* the NECT scan must be a NECT scan from the brain;
* the NECT scan must contain the entire brain
* the patient should have at least one of the following risk factors for developing a brain aneurysm

  * patient is female
  * patient has a family history of brain aneurysms
  * patient is 40 years or older
  * patient has or is treated for a high blood pressure
  * patient actively smokes cigarettes at time of inclusion
* a first informed consent form must be signed before brain NECT scans can be transferred to Robovision
* a second signed written informed consent must be obtained before follow-up data will be gathered, if applicable.

Exclusion Criteria:

- There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Verify the opportunistic screening potential of the AI software for detection of brain UIA on routinely performed brain NECT scans in a prospective setting | an average of 1 month after subject enrolment

SECONDARY OUTCOMES:
Verify the percentage of patients that underwent treatment(s) of the UIA after detection of the possible UIA by the AI software, confirmation of possible UIA by the radiologist, and definitive diagnosis of the UIA, by review of the EPD. | Through study completion, an average of 5 years.
Measure the health-related quality of life of patients by completion of the EQ-5D-5L questionnaire. | From start patient recruitment until 1 month after last patient signed ICF. Questionnaire to be completed 1 months after signing ICF.
Verify patients' complications by review of the EPD after 5 years | 5 years after patient enrolment.
  Patient outcomes measured 5 years after end of enrolment (Q4 2030) including whether or not the patient received complications related to the (non-)treated brain aneurysm, died, and/or whether the aneurysm has ruptured. Complications of ruptured brain aneurysms and subsequent subarachnoid hemorraghe can include, but are not limited to, cerebral vasospasm, hydrocephalus, hyponatremia, seizures, stroke, (permanent) brain damage, coma, and/or death.

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg - campus Sint-Jan, Genk
  - AZ Groeninge, Kortrijk
  - Ziekenhuis Oost-Limburg - campus Maas en Kempen, Maaseik

IPD SHARING:
Plan to Share IPD: No